CLINICAL TRIAL: NCT05770843
Title: Work Ability-Productivity Among Clinical Health Workers Endometriosis Study (Work ACHES): Protocol
Brief Title: Work Ability-Productivity Among Clinical Health Workers Endometriosis Study
Acronym: Work ACHES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Birkbeck, University of London (Other)
Responsible Party: Principal Investigator, Krystle Thomas Vedat, Doctoral student, Birkbeck, University of London
Other Study IDs: 50727
Record Dates: First submitted 2023-03-04; First posted 2023-03-16 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Endometriosis
Keywords: Work Ability; Work Productivity; Pain; Clinical Health Workers; Nurses; Doctors
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A qualitative multicentre study protocol. The prospective research explores clinical health workers with a diagnosis of endometriosis, experiencing regular pain and their perceptions of work ability-productivity.

DETAILED DESCRIPTION:
Endometriosis has a significant impact on women at work physically, psychologically, and socially. Notably, pain is the most common reported concern, and considerably reduces work ability and productivity. However, previous research has principally focused on general workers, discounting the varied nature of work roles. Health workers appear to have an increased occupational risk of developing the condition, when compared with other shift workers and the general working population. Taking these findings into account, the prospective WORK ACHES study explores the relationship between clinical health workers' regular endometriosis pain, and their perceptions of work ability-productivity during such events.

This multicentre qualitative study will invite employees with a diagnosis of endometriosis and working in clinical settings, to participate in the study. Recruitment will be carried out through study posters displayed in staff areas and occupational health departments, as well as snowballing methods. Semi-structured interviews will take place via Microsoft Teams to discuss participants' experiences of endometriosis pain at work and their work ability-productivity while symptomatic. Thematic analysis will be performed to interpret the data.

The study has sought ethical approval from Birkbeck University of London's ethics Committee, the Integrated Research Application System and the Health Research Authority. Following the completion of the study, a summary of findings will be shared with participants and agreed hospitals. The full study report will also be disseminated to all parties involved and accessed through the University of London's library thesis collection and published in relevant specialty journals.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18-65 years.
* Employed working within a clinical setting health role.
* English speaking.
* Currently working full or part time hours.
* Diagnosis of endometriosis (as reported by participant, as medical records will not be accessed for the purpose of this study).
* Experiences regular endometriosis associated pain.

Exclusion Criteria:

* Painful comorbidities.
* Unemployed women.
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Clinical health workers with a diagnosis of endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Perception of work ability-productivity during endometriosis associated pain | Up to 45 minutes
  Semi-structured interviews will be used to examine clinical health workers' perceived work ability-productivity during episodes of endometriosis associated pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Birkbeck, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No